CLINICAL TRIAL: NCT07368140
Title: Electrical Vestibular Stimulation as a Novel Neuromodulation Therapy for Vestibular Migraine: a Pilot Randomized Controlled Trial
Brief Title: Exploring Mild Electrical Vestibular Stimulation as a New Treatment for Dizziness and Migraine Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Neursantys Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB25-1327
Record Dates: First submitted 2025-11-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Vestibular Migraine
Keywords: Electrical Vestibular Stimulation; Galvanic Vestibular Stimulation; Vestibular Migraine; Vertigo; Dizziness; Balance and gait; Inertial Measurement Units; Motion sensitivity; Posturography; Neuromodulation
MeSH Terms: conditions — Vertigo; Dizziness

STUDY DESIGN:
Intervention Model Description: Two-arm, 1:1 randomized, parallel group design comparing active subthreshold stochastic electrical vestibular stimulation (EVS) to sham EVS, delivered across 6 sessions over 2 weeks, with symptom diaries and sensor-based balance and gait assessments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active subthreshold stochastic electrical vestibular stimulation (Experimental): Participants randomized to the active arm will receive subthreshold wideband stochastic electrical vestibular stimulation delivered via surface electrodes placed over the mastoid region and upper neck. Stimulation will be administered while seated in six sessions over two weeks. Each session will consist of two 20 minute stimulation blocks separated by a 5 minute rest. The current waveform will be a low amplitude stochastic signal (±0.35 mA) adjusted to remain below the threshold for overt vestibular sensations while providing continuous vestibular afferent input. Participants will be free to rest, read, or use personal devices during stimulation.
  Interventions: Device: Electrical Vestibular Stimulation
- Sham electrical vestibular stimulation (Sham Comparator): Participants randomized to the sham arm will undergo identical preparation, electrode placement, and scheduling as the active group, including six seated sessions over two weeks with two 20 minute blocks and a 5 minute rest per session. At the start of each block, the stimulator will briefly ramp up to a low current to mimic the sensation of active stimulation, then be reduced to zero current for the remainder of the session, while device indicators remain active. No therapeutic level vestibular stimulation will be delivered.
  Interventions: Device: Electrical Vestibular Stimulation Sham

INTERVENTIONS:
Device: Electrical Vestibular Stimulation — Subthreshold stochastic electrical vestibular stimulation delivered with a dual-channel isolated constant-current stimulator (Neursantys Inc.). Four-electrode mastoid-C4 montage; wideband stochastic current (0.001-300 Hz), ±0.35 mA (0.70 mA peak-to-peak), output sampled at 5 kHz. Two 20-minute seated stimulation blocks per session. Generates vestibular afferent activation while remaining below perceptual thresholds.
  Other Names: Galvanic Vestibular Stimulation
  Arms: Active subthreshold stochastic electrical vestibular stimulation
Device: Electrical Vestibular Stimulation Sham — Identical electrode placement and device setup as active electrical vestibular stimulation. Device ramps briefly, then delivers zero current for the remainder of the two 20-minute blocks. Device lights remain active to maintain masking; no vestibular stimulation is delivered after the ramp.
  Arms: Sham electrical vestibular stimulation

SUMMARY:
Vestibular migraine is a common cause of repeated dizziness, imbalance, and headaches that affects about three percent of Canadians. Many people do not find relief from current medications, leaving them with long term problems in balance and daily function. This study will test a new, non drug based treatment called electrical vestibular stimulation (EVS). EVS delivers gentle, safe electrical signals behind the ears to activate the brain's vestibular pathways.

Fifty adults with vestibular migraine will take part. Half will receive real stimulation, and half will receive a sham (placebo) treatment. Each participant will attend six sessions over two weeks. Around the treatment period, they will record dizziness and migraine symptoms in a daily diary and complete questionnaires and balance tests using motion sensors.

The main goal is to determine whether EVS can be delivered safely and comfortably in adults with vestibular migraine and whether participants can complete the sessions and assessments as planned. Results will also show whether symptoms or balance improve, providing essential information to design a larger clinical trial and, ultimately, develop new, accessible treatments for dizziness and migraine.

DETAILED DESCRIPTION:
Vestibular migraine (VM) is a neurological disorder in which recurrent vestibular symptoms such as vertigo, dizziness, and imbalance occur in association with migraine features. VM can produce persistent motion sensitivity, activity restriction, and functional impairment, and many individuals report incomplete relief of dizziness or imbalance with current pharmacologic strategies. Proposed mechanisms implicate altered multisensory integration across vestibular and migraine-related nociceptive networks, including abnormal brainstem and thalamocortical processing, trigeminal vestibular interactions, neuropeptide mediated neuroinflammation, cortical spreading depression, and central sensitization. These features motivate evaluation of non drug neuromodulation approaches that target vestibular pathway excitability and integration.

Electrical vestibular stimulation (EVS) is a non invasive neuromodulation technique that applies low amplitude electrical current through surface electrodes positioned over the mastoid and upper cervical region to modulate vestibular afferent activity and downstream central vestibular processing. Stochastic "noisy" wideband waveforms can provide continuous vestibular afferent input while remaining below thresholds for overt vestibular reflexes when delivered at subthreshold intensities. Prior balance focused studies have delivered repeated subthreshold stochastic EVS without serious adverse events, supporting evaluation of EVS as a portable and scalable intervention for vestibular conditions. This study is designed as a pilot randomized sham controlled trial to evaluate the feasibility safety and tolerability of repeated EVS delivery in adults with a confirmed clinical diagnosis of VM and to generate preliminary estimates of symptom and functional change to inform the design of a future fully powered randomized controlled trial.

Approximately 50 adults with VM will be recruited through the Calgary Headache Assessment and Management Program and affiliated clinics. Following informed consent and completion of baseline assessments participants will be randomized in a one to one ratio to receive either active EVS or sham EVS using a pre specified allocation schedule. Where feasible randomization will be stratified by sex to promote balance between groups given known sex differences in VM prevalence and symptom expression. The study will use a quadruple masking such that participants, care providers administering stimulation, investigators, and outcome assessors will remain blinded to group assignment throughout the study. Allocation concealment will be maintained by separating roles between personnel responsible for intervention delivery and those conducting outcome assessments. Procedures for unblinding will be after the data has been cleaned and groups need to be separated for comparisons.

Participants will attend six stimulation sessions scheduled across a two week intervention period. Stimulation will be delivered while seated using a wideband noisy waveform at a subthreshold intensity intended to avoid overt vestibular sensations while providing continuous vestibular afferent input. Each visit will include two 20 minute stimulation bouts separated by a 5 minute rest period. Standardized electrode placement skin preparation and impedance checks will be performed at each visit to ensure consistency across sessions. Participants will be allowed to read, rest, or use personal electronic devices during stimulation. Investigators will document session timing adherence and any deviations from the protocol as well as participant reported sensations during and after stimulation.

Participants assigned to the sham condition will undergo identical electrode placement and session structure as the active group. At the beginning of each stimulation bout the device will briefly ramp to mimic cutaneous sensation associated with stimulation onset and will then deliver zero current for the remainder of the bout while maintaining device indicators. This approach preserves participant expectations, staff interaction, and visit structure while withholding therapeutic vestibular stimulation. Study personnel will follow identical scripted procedures and monitoring protocols for both groups to support masking integrity.

Safety and tolerability will be monitored throughout the study period. Investigators will document the onset, duration, severity, and perceived relatedness of all reported events. Criteria for pausing or discontinuing stimulation during a session will be applied if participants experience concerning symptoms. Adverse events will be summarized by frequency severity and relatedness to inform safety characterization and protocol refinement.

Study assessments will be conducted at baseline immediately following completion of the two week intervention period and approximately one month after the final stimulation session. At each assessment, visit participants will complete validated patient reported measures capturing vestibular migraine related symptom impact, migraine related disability dizziness, related functional burden balance confidence, and motion sensitivity susceptibility. Structured symptom provocation procedures relevant to visually and vestibular triggered symptoms will also be completed to characterize changes in symptom sensitivity over time. Objective evaluation of postural control and functional gait will be performed using wearable inertial measurement units (IMUs). IMUs placed on the head trunk and feet will capture kinematic data during quiet standing performed under systematically varied sensory conditions and during standardized functional mobility tasks. These measures will be complemented by computerized dynamic posturography to quantify sensory integration during stance. Standardized task instructions, sensor placement, and trial timing will be used across visits to support consistency and data quality.

To capture day to day variability typical of vestibular migraine and to evaluate the feasibility of longitudinal symptom monitoring participants will complete daily symptom diaries for 30 days before and 30 days after the two week stimulation period. Diaries will record vestibular episode characteristics migraine features perceived symptom severity sleep and medication use. Completion rates and patterns of missing data will be tracked to inform feasibility and to guide protocol optimization for future trials. Among participants who menstruate daily tracking of menstrual bleeding will be included to support exploratory evaluation of symptom patterning.

The primary focus of this pilot trial is feasibility and tolerability, including recruitment and retention adherence to the six session intervention and acceptability of the intervention and assessments. Clinical and functional outcomes will be analyzed using longitudinal approaches appropriate for repeated measures to estimate the direction and variability of change over time between stimulation and sham groups. Effect sizes and confidence intervals will be reported rather than definitive hypothesis testing to support sample size estimation and design refinement for a future definitive randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of VM, according to the ICHD-3 and Barany Society criteria.
* Experienced at least one vestibular migraine episode in the previous month.
* Ability to provide informed consent and comply with study requirements.
* Willingness to attend six EVS sessions over a two-week period and complete all required testing and diaries.
* Physical ability to stand unassisted for at least one minute and walk 25 feet without assistance.

Exclusion Criteria:

* Diagnosis of other vestibular disorders (e.g. benign paroxysmal positional vertigo, Meniere's disease, vestibular neuritis) that may confound results.
* History of seizure disorder, epilepsy, or unexplained loss of consciousness.
* Presence of implanted electronic medical devices, such as pacemakers or cochlear implants.
* Pregnancy or plans to become pregnant during study period.
* Use of vestibular suppressant or migraine prophylactic medications that cannot be paused or maintained at a stable dose during the two-week EVS intervention period. Acute use of rescue medications during a severe attack is permitted, however, participants who initiate new medication or undergo dose changes during the intervention window will be excluded from final analysis.
* Current medical, psychiatric, or neurological condition (other than VM) that could interfere with participation.
* Cognitive or language impairments that preclude understanding of instructions or valid completion of outcome measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Vestibular Migraine Patient Assessment Tool and Handicap Inventory (VM PATHI) score | Baseline (pre intervention) to one month after completion of the two week EVS/sham intervention.
  The VM PATHI is a validated questionnaire specific to vestibular migraine that assesses six categories of patient reported outcome measures. It is a 25-item questionnaire scoring from 0 (best) - 100 (worst). The primary efficacy analysis will compare change in VM PATHI total score from baseline to one month post intervention between the active stimulation and sham groups using linear mixed effects models adjusted for baseline score, age, and sex.
Session Adherence (feasibility of delivering six Stim/Sham sessions) | From first stimulation session to end of the two week intervention period
  Proportion of randomized participants who complete at least five of six planned electrical vestibular stimulation or sham sessions within 14 days. Feasibility will be considered acceptable if at least 80 percent of participants meet this criterion.
Diary completion rate | 30 days prior to first stimulation session through 30 days after the final stimulation session (total 60 days)
  Proportion of days with a completed daily vertigo/migraine symptom diary during the 60 day monitoring period. Feasibility will be evaluated by the percentage of participants who complete diaries on at least 80 percent of days.
EVS related adverse events (safety and tolerability) | From baseline visit through one month post intervention follow up.
  Number and severity of device related adverse events, including skin irritation, discomfort, headache worsening, or other unexpected symptoms, recorded at each visit using a standardized adverse event log. Events will be summarized as counts and proportions per group and classified by seriousness and relatedness to the study device.

SECONDARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) score | Baseline, immediately post intervention, and one month post intervention
  The DHI is a 25 item questionnaire assessing self perceived handicap due to dizziness. Total scores (0-100) will be compared across time and between active and sham groups to evaluate changes in dizziness related disability.
Change in Activities specific Balance Confidence (ABC) scale score | Baseline, immediately post intervention, and one month post intervention
  The ABC scale is a 16-item questionnaire that assesses confidence in maintaining balance during daily activities. Percentage scores (0-100 percent) will be used to assess changes in balance confidence over time and between groups.
Change in Migraine Disability Assessment (MIDAS) scores | Baseline and one month post intervention
  The MIDAS is a 5-item questionnaire that captures frequency of headaches that affect certain tasks over 3-months. Scores are tallied from 0 (best) to 21+ (worst), indicating severe disability. Scores will be compared between active and sham groups to estimate the effect of electrical vestibular stimulation on migraine related disability.
Change in Motion Sickness Susceptibility Questionnaire (MSSQ) scores | Baseline and one month post intervention
  The MSSQ is an 18-item questionnaire that assesses susceptibility to motion sickness from 0 (best) to 54 (best). Changes in this score will be compared between stimulation and sham groups.
Change in Vestibular Ocular Motor Screening (VOMS) symptom provocation scores | Baseline and immediately post intervention
  VOMS symptom ratings (headache, dizziness, nausea, fogginess; 0-10 scale) will be recorded at baseline and after each VOMS task. There are 7 tasks. Composite change scores will be compared between groups to assess EVS related changes in visual vestibular integration and symptom provocation.
Change in modified Motion Sensitivity Test (mMST) score | Baseline and immediately post intervention
  The mMST consists of 10 standardized head and body movements with movement intensity ratings used to calculate a motion sensitivity score on a scale from 0-10 (worst). The duration it takes for the participant to return back to baseline after the movement is recorded and converted to points. The total score is calculated from intensity of the movement plus the duration it takes to return to baseline averages across movements to produce a percentage score where 0% (best) and 100% (worst). Changes in mMST percentage scores from baseline to post intervention will be compared between groups.
Change in IMU derived postural sway metrics during standing balance tests | Baseline, immediately post intervention, and one month post intervention
  IMUs placed on the head, trunk, and feet will record acceleration during quiet standing under four modified CTSIB conditions (firm vs foam surface, eyes open vs closed). Sway metrics (e.g., phybrata power, root mean square sway amplitude, average sway velocity, sway pathlength) will be computed. Changes over time and between groups will be used to quantify EVS effects on postural stability.
Change in gait performance during 25-foot walking test | Baseline, immediately post intervention, and one month post intervention
  Inertial measurement unit based gait metrics (e.g., cadence, step length, step width variability, head stabilization, and speed) will be extracted from the 25-foot walk. Between group differences in change over time will be used to evaluate electrical vestibular stimulation related improvements in gait stability.
Change in gait performance on Timed Up and Go (TUG) | Baseline, immediately post intervention, and one month post intervention
  Inertial measurement unit based gait metrics (time-to-completion, speed, head stability) will be extracted during TUG. Between group differences in change over time will be used to evaluate electrical vestibular stimulation related improvements in gait stability.
Change in Sensory Organization Test (SOT) equilibrium and sensory ratios | Baseline, immediately post intervention, and one month post intervention
  The SOT will be completed on the NeuroCom which uses computerized dynamic posturography to evaluate standing balance under 6 conditions. Equilibrium scores are produced for each condition from 0 (worst) to 100 (best) based on center of pressure during balance tasks. Sensory ratios are calculated by dividing equilibriums scores of specific conditions. The equilibrium scores and sensory ratios will be compared among groups.

OTHER OUTCOMES:
Menstrual cycle phase tracking | Daily menstrual tracking for 30 days before and 30 days after the intervention
  Among menstruating participants, daily diary entries will record menstrual bleeding. Exploratory analyses will examine whether changes in primary outcomes differ by menstrual cycle phase (bleeding vs non bleeding days).

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, University of Calgary, Calgary, Alberta, Canada